CLINICAL TRIAL: NCT04023760
Title: Pharmacokinetics of Apixaban and Tacrolimus or Cyclosporine in Kidney and Lung Transplant Recipients
Brief Title: Drug Interaction Study of Apixaban With Cyclosporine or Tacrolimus in Transplant Recipients
Acronym: ACT-KLR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other); Lung Association of Saskatchewan (Unknown)
Responsible Party: Principal Investigator, Holly Mansell, Associate Professor, College of Pharmacy and Nutrition, University of Saskatchewan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 99861
Record Dates: First submitted 2019-06-28; First posted 2019-07-18 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Pharmacokinetics; Kidney Transplant; Lung Transplant
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Treatment group A: Cyclosporine in transplant recipients (Experimental): A single oral dose of 10 mg apixaban will be administered to kidney or lung transplant recipients stabilized on cyclosporine as part of their immunosuppressive regimen
  Interventions: Drug: Apixaban
- Cyclosporine in healthy subjects (Active Comparator): Results from Treatment group A will be compared to previously obtained data in healthy participants receiving a single dose of apixaban with a daily dose of 100 mg of cyclosporine at steady state concentration (Bashir et al. Clin Transl Sci. 2018 Jul 3. doi: 10.1111/cts.12580)
  Transplant recipients require continuous immunosuppression so it will not be possible to stop the cyclosporine or tacrolimus to serve as a control. As such PK plasma time curves will be compared to data in healthy volunteers.
  Interventions: Drug: Apixaban
- Treatment group B: Tacrolimus in transplant recipients (Experimental): A single oral dose of 10 mg apixaban will be administered to kidney or lung transplant recipients stabilized on tacrolimus as part of their immunosuppressive regimen
  Interventions: Drug: Apixaban
- Tacrolimus in healthy subjects (Active Comparator): Results from Treatment group B will be compared to previously obtained data in healthy participants receiving a single dose of apixaban with a daily dose of 100 mg of tacrolimus at steady state concentration (Bashir et al. Clin Transl Sci. 2018 Jul 3. doi: 10.1111/cts.12580)
  Transplant recipients require continuous immunosuppression so it will not be possible to stop the cyclosporine or tacrolimus to serve as a control. As such PK plasma time curves will be compared to data in healthy volunteers.
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Study subjects given a single-dose of apixaban 10 mg.
  Other Names: Eliquis

SUMMARY:
This study aims to evaluate the pharmacokinetics (PK) of apixaban in kidney and lung transplant recipients stabilized on either cyclosporine or tacrolimus as part of their immunosuppressive therapy.

DETAILED DESCRIPTION:
Solid organ transplantation is a lifesaving option for many patients with end-stage organ disease. After transplant surgery, patients must take immunosuppressive therapy, which carries significant risk for drug-drug interactions and adverse medication-related events.

Transplant recipients are at an increased risk for co-morbidities traditionally managed with warfarin, such as venous thromboembolism and atrial fibrillation. Apixaban has the potential to provide safer and more effective treatment, without additional monitoring of the INR, but it has not been studied in conjunction with anti-rejection agents in this population. Apixaban is metabolized by CYP3A4 and P-gp and BCRP transporters. As part of their immunosuppressive therapy, solid organ transplant recipients are maintained on calcineurin inhibitors, which are weak CYP3A4 as well as potent P-gp and BCRP inhibitors. A study was recently undertaken to evaluate the potential drug-drug interaction between cyclosporine or tacrolimus and apixaban in healthy subjects (ClinicalTrials.gov Identifier: NCT03083782) . The results indicated that the change in apixaban exposure was not clinically relevant.

PK studies in healthy volunteers are a first step for determining the nature and extent of potential drug-drug interactions. However, follow-up studies in the actual patient populations are essential for ensuring safety and tolerability, and providing clinicians the confidence to use these combinations. The purpose of this study is to confirm the pharmacokinetic characteristics and safety of apixaban in combination with tacrolimus and cyclosporine in stable kidney and lung transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Kidney or lung transplant patients followed as outpatients who are currently stabilized on immunosuppressive therapy with tacrolimus or cyclosporine
* Age 18 or older
* At least six months after transplantation
* Lack of transplant rejection within the last 12 weeks
* Creatinine clearance at least above 15ml/min as calculated by Cockroft-Gault formula
* Negative urine pregnancy test for female patients of childbearing potential
* Consent to the study
* Be a nonsmoker for at least approximately 6 months prior to the study
* Have a prothrombin time (PT) and activated partial thromboplastin time (PTT) level below the upper limit of normal
* Have a hemoglobin level of above at least 80g/L
* Be willing to refrain from the use of anticoagulants and antiplatelet medications including aspirin and non-steroidal anti-inflammatory drugs (NSAIDs) for two weeks prior and during the entire period of study participation
* Be willing to avoid drinking grapefruit juice or consuming natural health products for two weeks prior and during the study period
* Be willing to avoid alcohol and cannabis for 48 hours before the study and for the entire duration of the study
* Be willing to comply with trial restrictions
* Be deemed safe to participate by the study physician

Exclusion Criteria:

* Patients on antiplatelet therapy for any cardiovascular treatment (such as clopidogrel, prasugrel, ticagrelor). Patients on prophylactic aspirin will be eligible otherwise.
* Patients not receiving tacrolimus or cyclosporine
* A history of an anaphylactic or severe systemic reactions to apixaban
* Any form of substance abuse or major untreated psychiatric disorder
* Pregnancy or lactation
* Tacrolimus or cyclosporine changes within the last two weeks
* Receiving concurrent therapy with warfarin, or are taking medications known to be strong inhibitors of both cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp) such as azole-antimycotics antifungals (e.g., ketoconazole, voriconazole.)
* Has congenitial or acquired coagulation disorders
* Has moderate or severe hepatic disease or other clinically relevant bleeding risk
* Use of any drugs or products which at the discretion of the investigator would increase bleeding risk
* Has any unstable medical condition that could interfere with the study
* Is considered inappropriate for participation by the investigator for any reason
* Clinically significant active bleeding, including gastrointestinal bleeding
* Lesions or conditions at increased risk of clinically significant bleeding, e.g., recent cerebral infarction (ischemic or hemorrhagic), active peptic ulcer disease with recent bleeding, patients with spontaneous or acquired impairment of hemostasis
* Patients who donate blood within 56 days of participating in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Apixaban area under the plasma concentration curve between 0 and 72 hours (AUC(0-72)). | Days 1-3
  Blood samples for Apixaban pharmacokinetics will be collected prior to apixaban administration at 0H, and then at 1, 2, 3, 4, 6, 12, 24, 48 and, 72 hours in each treatment arm
Apixaban peak plasma concentration (Cmax) | Days 1-3
  Blood samples for Apixaban pharmacokinetics will be collected prior to apixaban administration at 0H, and then at 1, 2, 3, 4, 6, 12, 24, 48 and, 72 hours in each treatment arm.

SECONDARY OUTCOMES:
Safety and tolerability of Apixaban when co-administered with cyclosporine assessed by capturing incidence of adverse events | Days 1-4
  Number of participants who experience an adverse events based on the results of laboratory safety tests and the results of vital sign measurements, physical examinations, and clinical laboratory tests
Safety and tolerability of Apixaban when co-administered with tacrolimus assessed by capturing incidence of adverse events | Days 1-4
  Number of participants who experience an adverse events based on the results of laboratory safety tests and the results of vital sign measurements, physical examinations, and clinical laboratory tests

OTHER OUTCOMES:
Differences in area under the plasma concentration curve between 0 and 72 hours AUC (0-72)) in kidney and lung transplant recipients | Days 1-3
  Blood samples for Apixaban pharmacokinetics will be collected prior to apixaban administration at 0H, and then at 1, 2, 3, 4, 6, 12, 24, 48 and, 72 hours in each treatment arm
Differences in peak plasma concentration (Cmax) hours between kidney and lung transplant recipients | Days 1-3
  Blood samples for Apixaban pharmacokinetics will be collected prior to apixaban administration at 0H, and then at 1, 2, 3, 4, 6, 12, 24, 48 and, 72 hours in each treatment arm
Differences in area under the plasma concentration curve between 0 and 72 hours AUC(0-72)) between transplant recipients and healthy subjects | Days 1-3
  Blood samples for Apixaban pharmacokinetics will be collected prior to apixaban administration at 0H, and then at 1, 2, 3, 4, 6, 12, 24, 48 and, 72 hours in each treatment arm
Differences in peak plasma concentration (Cmax) hours between transplant recipients and healthy subjects | Days 1-3
  Blood samples for Apixaban pharmacokinetics will be collected prior to apixaban administration at 0H, and then at 1, 2, 3, 4, 6, 12, 24, 48 and, 72 hours in each treatment arm

CONTACTS AND LOCATIONS:
Locations (1):
- Saskatchewan Health Authority, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bashir B, Stickle DF, Chervoneva I, Kraft WK. Drug-Drug Interaction Study of Apixaban with Cyclosporine and Tacrolimus in Healthy Volunteers. Clin Transl Sci. 2018 Nov;11(6):590-596. doi: 10.1111/cts.12580. Epub 2018 Jul 27. PMID 29972633
- [Derived] Mansell H, Shoker A, Alcorn J, Fenton ME, Tam JS, Semchuk W, Bashir B, Kraft WK, Yao S, Douketis JD. Pharmacokinetics of apixaban and tacrolimus or cyclosporine in kidney and lung transplant recipients. Clin Transl Sci. 2022 Jul;15(7):1687-1697. doi: 10.1111/cts.13284. Epub 2022 May 2. PMID 35439353